CLINICAL TRIAL: NCT03910062
Title: Lower Limb Surveillance During VA-ECLS: Evaluation of Angiography Through the Reperfusion Cannula at VA-ECMO Implantation and of Near Infrared Spectroscopy (NIRS) Monitoring
Brief Title: Lower Limb Surveillance During VA-ECLS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2018/MIRECMO-KOSZUTSKI/YB
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2020-03

CONDITIONS: Cardiogenic Shock; Cardiac Arrest; Lower Limb Ischemia
Keywords: VA-ECMO; VA-ECLS; Near-Infrared Spectroscopy (NIRS)
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VA ECMO: Patients under VA-ECMO with a femoral reperfusion cannula.
  Interventions: Procedure: Lower limb angiography via the reperfusion cannula and NIRS monitoring

INTERVENTIONS:
Procedure: Lower limb angiography via the reperfusion cannula and NIRS monitoring — Data collection only (lower limb angiography, lower limbs NIRS values).

SUMMARY:
Temporary cardiac support by VA-ECLS can lead to lower limb ischemia. The aim of this study is to evaluate a multi-modal strategy (physical examination, NIRS monitoring and angiography through the reperfusion canula) of lower limb surveillance.

DETAILED DESCRIPTION:
VA ECLS is used as a temporary circulatory support during cardiogenic shock and refractory cardiac arrest. Complications of VA ECLS include hemorrhagic, infectious and ischemic events. VA ECLS requires arterial and venous canules which are frequently positioned in the femoral artery and vein, which carries the risk of lower limb ischemia due to retrograde flow and obstruction of the femoral artery lumen. VA ischemia during VA ECLS is frequent (11-52%) and requires the use of reperfusion canula in the femoral common artery on VA ECLS implantation in a primary prevention strategy, before lower limb ischemia occurs. Even with this strategy, lower limb ischemia can occur due to arterial thrombosis, arterial spasm or insufficient blood flow through the reperfusion canula. Lower limb complications are prevented by monitoring of regional oxygen saturation, control of the reperfusion canula position (ultrasound, angiography) and rapid management when lower limb ischemia is suspected. There are no clear recommendations regarding prevention of lower limb complications during VA ECLS and arterial angiography has been described to diagnose ischemic events and evaluate the effectiveness of an intervention such as injection of vasodilators. This study is a prospective evaluation of a strategy to prevent lower limb complications during VA ECLS with a systematic arterial angiography on VA ECLS implantation and when lower limb ischemia is suspected (regional oxygen tissue saturation <50% or a differential >15% between both lower limbs) in addition to continuous NIRS monitoring of lower limbs during VA ECLS.

ELIGIBILITY:
Inclusion Criteria:

* Temporary circulatory support with VA ECLS
* Age > 18 years

Exclusion Criteria:

* Pregnancy
* History of iodinated contrast allergy
* History of lower limb amputation above the ankle
* Lower limb ischemia before starting of VA-ECLS
* Femoro-axillary VA-ECLS
* Absence of the lower limb reperfusion canula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under Temporary Cardiac Support with VA-ECLS
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Severe limb ischemia | 60 days
  Ischemia leading to surgical intervention, functional sequelae, necrosis of the extremities or compartment syndrome

SECONDARY OUTCOMES:
Mortality | 28 days and 60 days
  Mortality rate
Incidence of ischemia of the lower limb during ICU stay | 2 months
  StO2 < 50% during 4 consecutive minutes AND/OR StO2 differential > 15% during ICU stay
Incidence of renal replacement therapy during ICU stay | 2 months
  Number of patients who underwent renal replacement therapy
Duration of ICU stay | 60 days
  Number of days in the ICU
Duration of hospital stay | 60 days
  Number of days in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Koszutski, Dr, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koszutski M, Mattei M, Maureira JP, Kimmoun A, Levy B. Assessment of bedside lower limb angiography combined with continuous NIRS monitoring for the detection of lower limb complications of VA-ECMO: an observational monocentric study. Crit Care. 2021 Jul 31;25(1):270. doi: 10.1186/s13054-021-03703-5. PMID 34332620